CLINICAL TRIAL: NCT02332122
Title: Detection of Aspergillus Fumigatus and Sensitization in COPD Patients With Bronchiectasis vs COPD Patients Without Bronchiectasis
Brief Title: Detection of Aspergillus Fumigatus and Sensitization in COPD Patients With Bronchiectasis vs Without Bronchiectasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wim Janssens (Other)
Responsible Party: Sponsor-Investigator, Wim Janssens, MD. PhD, KU Leuven
Organization: KU Leuven (Other)
Other Study IDs: S57222
Record Dates: First submitted 2015-01-05; First posted 2015-01-06 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Aspergillus fumigatus; Bronchiectasis; Sensitization; Vitamin D
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiectasis | interventions — Patch Tests; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum sample obtained through induction
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- COPD patients with bronchiectasis: All patients will receive standard therapy for AECOPD.
  Additional for this study are:
  Sputum induction, Skin prick test, Questionnaires
  Interventions: Procedure: Sputum induction; Procedure: Skin prick test; Other: Questionnaires
- COPD patients without bronchiectasis: All patients will receive standard therapy for AECOPD.
  Additional for this study are:
  Sputum induction, Skin prick test, Questionnaires
  Interventions: Procedure: Sputum induction; Procedure: Skin prick test; Other: Questionnaires

INTERVENTIONS:
Procedure: Sputum induction — Patients will have to puff 200µg of salbutamol (metered-dose inhaler with spacer device). After 10 minutes FEV1 will be measured with MIR spirobank. If FEV1 is >= 30% we can safely proceed with sputum induction. An ultrasonic nebulizer will be used to induce sputum. 4% sodiumchloride will be inhaled. Induction will be performed at 5-min intervals until a sample of good quality is obtained. Sodiumchloride of 5% will be used if no good sample is obtained after two intervals with the 4% solution. Maximal time of induction will be 20 minutes. Subjects will spit saliva into one container and rinse the mouth thoroughly with water before coughing sputum into another sterile container. Samples will be refrigerated at 4°C and processed within 24 hours of collection.
Procedure: Skin prick test — Skin Prick Test is a reliable method to diagnose IgE-mediated allergic disease. It is minimally invasive and results are immediately available. Interpretation utilizes the presence and degree of cutaneous reactivity as a surrogate marker for sensitization. A positive control, a negative control and Aspergillus fumigatus will be tested. Location will be Protocol version 1 3/11/2014 marked on the volar aspect of the forearm and drops of each solution will be placed (>= 2cm between drops). A single-head metal lancet will be pressed through the drop of allergen extract and held against the skin for at least 1 second. A new lancet will be utilized for each drop. A wheal diameter of >= 3mm is a positive result.
Other: Questionnaires — MRC: Medical Research Council Scale CAT: COPD Assessment Test SGRQ: Saint George's respiratory questionnaire

SUMMARY:
A single center case-control study with 100 COPD patients will be organized to compare patients with and without bronchiectasis with regard to the presence of Aspergillus in sputum samples, Aspergillus sensitization and vitamin D. Induced sputum samples will be optimized for culture, Aspergillus galatomannan analysis and RT-PCR.

This study is part of a larger project in which we assume that chronic respiratory infection by Aspergillus fumigatus and the accompanying immune response play an important role in the development of bronchiectasis in COPD. We suspect that this mechanism is controlled by vitamin D and it fails by suppression of the vitamin D receptor by Aspergillus fumigatus.

The present study is designed by the Laboratory of pneumology and will be conducted in collaboration with the Laboratory of clinical bacteriology and mycology of the Catholic University of Leuven.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of COPD by medical doctor (based on clinical history or pulmonary function test)
* Smoking history of at least 10 pack-years
* CT Thorax available for assessment of bronchiectasis
* FEV1 >= 30%

Exclusion Criteria:

* Mechanical or non-invasive ventilation
* Other main respiratory diagnosis other than COPD
* Active mycobacterial disease
* Immunosuppression other than steroids
* Active cancer treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present in the emergency department with an acute COPD exacerbation (as defined by GOLD executive summary) requiring hospitalization are eligible for this study. Patients should have an established diagnosis of COPD (based on clinical history or pulmonary function test). They will be recruited during their hospital stay in the University Hospital of Leuven.
  Additionally, we will include 20 patients with COPD (10 with bronchiectasis versus 10 without) in stable state during their outpatient visits.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Bronchiectasis | immediate

SECONDARY OUTCOMES:
Vitamin D | immediate
Prevalence of Aspergillus sensitization | max 12weeks
Prevalence of Aspergillus isolation in sputum | max 12weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wim Janssens, MD. PhD, Principal Investigator — KU Leuven - UZ Leuven
Locations (1):
- UZ Gasthuisberg, Leuven, Flanders, Belgium